CLINICAL TRIAL: NCT06299696
Title: A Phase 1, Open-label Taste Assessment Study of Vanzacaftor/Tezacaftor/Deutivacaftor in Healthy Adult Panelists
Brief Title: A Study of Vanzacaftor/Tezacaftor/Deutivacaftor (VNZ/TEZ/D-IVA) in Healthy Adult Panelists
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vertex Pharmaceuticals Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: VX23-121-011
Record Dates: First submitted 2024-02-29; First posted 2024-03-08 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis | interventions — deutivacaftor, tezacaftor , vanzacaftor

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- VNZ/TEZ/D-IVA (Experimental): Participants will be given VNZ/TEZ/D-IVA FDC to retain in their mouths for approximately 10 seconds and then expectorated.
  Interventions: Drug: VNZ/TEZ/D-IVA

INTERVENTIONS:
Drug: VNZ/TEZ/D-IVA — FDC granules for oral administration
  Other Names: VX-121/VX-661/CTP-656; VX-121/VX-661/VX-561; Vanzacaftor/tezacaftor/deutivacaftor

SUMMARY:
The purpose of this study is to evaluate the flavor (basic tastes, aroma, texture, mouthfeel) of VNZ/TEZ/D-IVA fixed dose combination (FDC) granules.

DETAILED DESCRIPTION:
This clinical trial information was submitted voluntarily under the applicable law and, therefore, certain submission deadlines may not apply. (That is, clinical trial information for this applicable clinical trial was submitted under section 402(j)(4) (A) of the Public Health Service Act and 42 CFR 11.60 and is not subject to the deadlines established by sections 402(j)(2) and (3) of the Public Health Service Act or 42 CFR 11.24 and 11.44.).

ELIGIBILITY:
Key Inclusion Criteria:

* Panelists are trained to detect, identify, recognize, and accurately describe different taste elements and flavor combinations.

Key Exclusion Criteria:

* History of any illness or clinical condition that, in the opinion of the investigator, might confound the results of the study or pose an additional risk to the participant.
* Sensitivity to VNZ, TEZ, or D-IVA.
* Pregnant, nursing, or planning to become pregnant during the study

Other protocol defined Inclusion/Exclusion criteria may apply.

Ages: 25 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2024-03-26 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Flavor Assessment Based on Flavor Profile Method of Descriptive Sensory Analysis per American Society for Testing and Material (ASTM) Approved Sensory Evaluation Method | Periodic Intervals up to 30 minutes post oral administration

CONTACTS AND LOCATIONS:
Locations (1):
- Site 001, Woburn, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
Details on Vertex data sharing criteria and process for requesting access can be found at: https://www.vrtx.com/independent-research/clinical-trial-data-sharing